CLINICAL TRIAL: NCT02806258
Title: Comparing Sequential Neoadjuvant Treatment Including Chemotherapy and Accelerated Radiation Focused to the Tumor Bed vs Neoadjuvant Chemotherapy Alone, for Triple Negative Locally Advanced Breast Cancers and Luminal B Proliferating, Inaccessible to a Conservative Surgery the Outset
Brief Title: Comparing Sequential Neoadjuvant Treatment Including Chemotherapy and Accelerated Radiation Focused to the Tumor Bed vs Neoadjuvant Chemotherapy Alone
Acronym: Néo-APBI-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC14.454
Record Dates: First submitted 2016-04-06; First posted 2016-06-20 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Radiation Therapy, Breast Cancer, Sequential Partial Breast Irradiation; Intermediate and High-risk Luminal and Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): 6-8 cycles of Primary systemic therapy using anthracycline and/or taxane based regimens, according to their physician's preference and center policy
  Interventions: Drug: Chemotherapy
- Arm B (Experimental): The patients will receive 3D conformal or other modality (eg IMRT, VMAT) APBI during their PST sequence. APBI will be planned sequentially between the Primary systemic therapy cycles, 2 weeks after the 3rd/6 or the 4th/8 cycle of PST.
  Interventions: Radiation: Accelerated partial breast irradiation; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Accelerated partial breast irradiation — To date, there is no report on external beam APBI associated with CT in the neoadjuvant setting.In the NeoAPBI 01 trial, the objective is to demonstrate the efficacy of combined APBI and CT administered sequentially in patients with intermediate ad high risk BC. The hypothesis is that combined PST-sequential APBI may increase the rate of pCR, breast conservation and survival without additional toxicity, as seen with WBI.
  Arms: Arm B
Drug: Chemotherapy — minimum of six cycles of PST using anthracycline and/or taxane based regimens

SUMMARY:
In the NeoAPBI 01 trial, the objective is to demonstrate the efficacy of combined APBI and CT administered sequentially in patients with intermediate ad high risk BC. The hypothesis is that combined PST-sequential APBI may increase the rate of pCR, breast conservation and survival without additional toxicity, as seen with WBI

DETAILED DESCRIPTION:
Phase I:

The total APBI dose is set to level I at 20 Gy (in 10 fractions over 5 days; n=5) and then level II at 24 Gy (in 12 fractions over 6 days) delivered to the tumor using two fractions/day of 2 Gy spaced by at least 6 hours. The biological effective dose (BED) is 32 Gy and 47 Gy for alpha/beta of 10 and 3.5, respectively. As compared to the standard fractionation of 2 Gy/fraction the BED is 26.8 Gy and 30 Gy for the 2 values of alpha/beta.

In case of the impossibility to deliver two fractions/day, patients should be treated using a single fraction of 3.125 Gy/day up to 8 fractions (total dose of 25 Gy). The BED is 32.8 Gy and 47.3 Gy for alpha/beta of 10 and 3.5, respectively. As compared to the standard fractionation of 2 Gy/fraction the BED is 27.3 Gy and 30.1 Gy for the 2 values of alpha/beta.

In both schemes, 95% of the prescribed dose should be delivered in at least 90% of the PTV.

All patients who undergo BCS after the end of PST-APBI will receive postoperative WBI (+/- nodal areas) delivering a total dose of 45-50 Gy using standard fractionation (1.8 or 2 Gy) or hypofractionated schedules using > 15 fractions in 3 weeks. Technique and boost delivery will be left at the investigator's discretion and local policy. Patients who had TM should also receive PMRT if indicated delivering 45-50.4 Gy using standard fractionation (1.8 or 2 Gy). If the patient did not complete a full course of PST prior to surgery, CT will be given prior to or immediately following postoperative RT depending on the institutional protocol. Other post-operative treatments will be at the investigator's discretion. Adjuvant hormonal treatment will be administered to HR+ patients.

Phase II:

This is a phase II randomized study designed for patients with newly diagnosed intermediate and high risk non-metastatic BC who are candidates for a minimum of six cycles of PST using anthracycline and/or taxane based regimens, who desire BCS but are not eligible due to tumor/breast ratio. All patients will have a clip in the tumor bed before or after the first 1-2 cycles of PST.

Eligible patients who have consented to participate in the study will be randomized to treatment Arm A or B:

Arm A: 6-8 cycles of PST using anthracycline and/or taxane based regimens, according to their physician's preference and center policy.

Arm B: The patients will receive 3D conformal or other modality (eg IMRT, VMAT) APBI during their PST sequence. APBI will be planned sequentially between the PST cycles, 2 weeks after the 3rd/6 or the 4th/8 cycle of PST.

For the purpose of quality of the target volume definition, it is mandatory to make a planning CT-scan in treatment position before the initiation of chemotherapy. MRI or US fusion with CT scan images can increase target volume definition and should be used if necessary. For all patients, treatment planning should be made on a planning CT-scan shortly preceding the initiation of radiation therapy to take possible tumor shrinkage and breast shape changes into account.

The CTV is defined as GTV + 1cm. The margin to the PTV depends on the measurements of the center and thereby the positioning and verification techniques. If this is not known, PTV should be defined as CTV + 1 cm around. The PTV should be used for beam shaping while for dose evaluation and calculation a PTVeval will be defined as PTV excluding the skin + 5 mm and the thoracic wall (ribs and intercostal muscles). IMRT should not be used in the protocol. The PTVeval should not exceed 40% of the total breast volume.

Study Arms:

All patients must undergo surgery even in cases of clinical complete response. Surgery will be scheduled 4 to 6 weeks from the last day of PST.

Modified radical mastectomy is indicated in case of limited clinical response, or progressive disease, or if tumor size/breast size does not permit BCS. The decision should be based on US or MRI confirmation of the response. Post TM radiation therapy should be applied according to the center's guidelines. High risk patients should receive nodal radiotherapy policy.

All patients who undergo BCS after the end of PST-APBI, will receive postoperative RT. This will consist of WBI (+/- nodal areas) to a total dose of 45-50 Gy using standard fractionation (1.8 or 2 Gy) or hypofractionated schedules using > 15 fractions in 3 weeks. Technique and boost delivery will be left at the investigator's discretion and local policy. Patients who had TM should also receive PMRT, 45-50.4 Gy using standard fractionation (1.8 or 2 Gy). If the patient did not complete a full course of PST prior to surgery, CT will be given prior to or immediately following postoperative RT depending on the institutional protocol. Other post-operative treatments will be at the investigator's discretion. Adjuvant hormonal treatment will be administered to HR+ patients.

Standard protocol:

The patients randomized to the standard treatment arm will receive a minimum of 6-8 cycles of PST using an anthracycline and/or taxane based regimen. Surgery will consist of BCS or TM according to clinical response and tumor/breast volume ratio obtained after PST. After surgery, the patients will receive standard RT to the whole breast (45-50.4 Gy in 25-28 fractions) or equivalent using hypofractionated schedule > 15 fractions in 3 weeks. RT technique and the addition of boost are left to the investigator decision according to institutional protocol. Adjuvant ET will be administered to HR+ patients after the end of radiotherapy during at least 5 years.

Auxiliary translational study Tumor core biopsies for translational studies and genetic analysis will be obtained at baseline and from the resected tumor at surgery following PST +/- APBI.

This study will focus on the prediction of pCR using cell metabolism, hypoxia and angiogenesis markers (Scottish Group). Another objective is to correlate these markers with the metabolic imaging for pCR prediction (Oscar Lambret Center, France).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Histologically confirmed invasive carcinoma of the breast
* Patient who desires breast conservation
* Tumor stage T1N1, T2-3 N0-1
* Operable BC for which an indication for CT is determined, including T1N1 and high risk T2-3 N0-1 tumors.
* Lobular and/or ductal invasive carcinoma
* Confirmation by imaging (standard +/- MRI) of unicentric and unilateral disease
* Luminal B (defined by hormone receptor positive and grade II-III (if available from core biopsy) and Ki67 ≥ 15% or by genomic analysis) and TNG subtypes
* HER2 negative
* No distant metastases
* No contraindication for PST with anthracycline and/or taxane based regimens
* Patients with no psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator with the aid of written information.

Exclusion Criteria:

* Patients considered too frail for CT whatever their age.
* Breast cancer clinical grade T4 and /or with major nodal involvement N2 (clinically, US, MRI or PET-CT).
* Lumpectomy is considered to be possible with an anticipated favourable cosmetic outcome considering the tumor size/breast size
* Multicentricity that would not allow BCS as confirmed by breast imaging
* Uni or bilateral inflammatory (T4d) BC
* Metastatic disease
* Other histology types: ciribriform or tubular or mucinous or epideroid carcinomas
* Her2 positive
* No signed consent to participate in the study
* Previous malignancy (except non melanoma skin cancer, thyroid carcinoma, non-invasive cancers outside the breast and patients with previous cancer in remission since more > 5 years)
* Patients with psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule
* Patients unwilling or unable to comply with the protocol (especially necessity to undergo breast surgery despite clinical complete response)
* Patients who have received any other investigational drugs within 30 days prior to the screening visit
* Pregnancy
* Active connective tissue disease involving the skin
* Patients with other concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2016-04-26 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
PCR rates | At the end of chemotherapy: up to 21 weeks
  Pathological complete response (pCR), defined by the absence of invasive residual primary tumor in the breast and lymph node.The primary objective of this study is to compare pCR rates after Primary Systemic Therapy (PST) plus APBI versus PST alone in patients with luminal and TNG BC prior to BC surgery.

SECONDARY OUTCOMES:
PCR 2 | At the end of chemotherapy: up to 21 weeks
  Breast and axilla pathological complete response rate (pCR2)
Breast conservation rate | Intraoperative
  Breast conservation rate
Acute and late toxicities | At the end of chemotherapy and after surgery and after radiotherapy: up to 30 weeks
  Acute and late toxicities (CTCAE v 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Gabelle Flandin, Dr, Principal Investigator — CHU Grenoble Alpes
Locations (6):
- France (6):
  - CHI Créteil, Créteil
  - CHU de Grenoble, Grenoble
  - AP-HP Henri mondor, Paris
  - CHU Avicenne, Paris
  - H. Hartmann Institute of Radiotherapy and Radiosurgery, Paris
  - Tenon hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] To NH, Gabelle-Flandin I, Luong TMH, Loganadane G, Ouidir N, Boukhobza C, Grellier N, Verry C, Thiolat A, Cohen JL, Radosevic-Robin N, Belkacemi Y. Pathologic Response to Neoadjuvant Sequential Chemoradiation Therapy in Locally Advanced Breast Cancer: Preliminary, Translational Results from the French Neo-APBI-01 Trial. Cancers (Basel). 2023 Mar 29;15(7):2030. doi: 10.3390/cancers15072030. PMID 37046691